CLINICAL TRIAL: NCT06305169
Title: Measuring the Negative Predictive Value and Specificity of Serum Biomarkers in Gastric Cancer Along With Creating a Predictive Model for the Identification of Patients That Need Urgent Endoscopy
Brief Title: Measuring the Negative Predictive Value and Specificity of Serum Biomarkers in Gastric Cancer
Status: Not yet recruiting | Type: Observational
Sponsor: Sandwell & West Birmingham Hospitals NHS Trust (Other)
Responsible Party: Principal Investigator, Nigel Trudgill, Consultant Gastroenterologist, Sandwell & West Birmingham Hospitals NHS Trust
Other Study IDs: 1.4
Record Dates: First submitted 2024-02-28; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Referrals to endoscopy via the 2 week wait cancer pathway for all indications other than dysphagia: This group will have their serum biomarkers measured by gastropanel a commercially available blood test, along with full blood count and complete a questionnaire.
  Interventions: Diagnostic Test: Gastropanel

INTERVENTIONS:
Diagnostic Test: Gastropanel — Gastropanel is a commercially available blood test which given serum levels of pepsinogen I and II and gastrin 17 along with helicobacter pylori infection status

SUMMARY:
Atrophic gastritis where the cells of the stomach lining change is the single most important precursor condition for gastric cancer. Helicobacter pylori a bacteria which causes infection in the stomach is the most important causative agent of inflammation of the stomach, and subsequent atrophic gastritis.

The difficulty with diagnosing patients with gastric cancer is that a lot of patients will suffer from heartburn and pain around the stomach, but very few of those will have gastric cancer. This makes it difficult for GPs to know who to refer for further testing as the current cancer referral criteria are very broad.

To reduce the need for invasive diagnostic methods such as endoscopy where a flexible tube with camera is inserted into the gullet and stomach via the mouth, a commercially available blood test (GastroPanel ®) designed to measure the levels of certain key stomach hormones to detect atrophic gastritis has been developed. It is extremely rare for gastric cancer to develop without there first being gastric atrophy.

A real word study is needed assess the performance of this blood test in a group of patients referred via an urgent cancer pathway for endoscopy in the UK. Scoring systems have been created to help us triage referrals to endoscopy in those with difficulty swallowing, but no similar score is available for those presenting with other upper abdominal symptoms. By using this blood test as well as collecting patient information we hope to create an improved referral criteria for those needing investigation for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

Patients referred for a 2 week wait cancer pathway endoscopy for the following indications Or Upper abdominal mass consistent with stomach cancer Or Stable upper gastrointestinal bleeding Or

Aged 55 and over with weight loss and any of the following:

* Upper abdominal pain
* Reflux
* Dyspepsia

Exclusion Criteria:

* Referrals for therapeutic OGD (e.g. polypectomy, feeding tube insertion)
* Previous gastro-duodenal surgery,
* Any co-morbidity that may impair ability to provide information or give valid consent (e.g. dementia, cerebral vascular disease)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will consist of those patients referred primarily from their general practice for a cancer pathway endoscopy at the study site.
Sampling Method: Non-Probability Sample
Enrollment: 440 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of the specificity and negative predictive value of serum biomarkers in gastric cancer | 12 months
  Gastric serum biomarkers measured by gastropanel will be measured in 400 patients who undergo endoscopy. The research team will measure the specificity and negative predictive value of gastropanel in excluding gastric cancer in patient enrolled into the study.

SECONDARY OUTCOMES:
Creating a scoring system for patients that warrant urgent endoscopy on the cancer pathway | 3 months
  By using the hormone levels detected in the gastropanel blood test along with a blood test to check for anaemia (low red blood count), patient questionnaire looking at symptoms and the patients medical background the research team will use logistic regression analysis to identify factors strongly associated with cancer diagnosis and derive a risk score.

CONTACTS AND LOCATIONS:
Locations (1):
- Sandwell General Hospital, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Anonymised aggregated data can be requested by other researchers